CLINICAL TRIAL: NCT03515486
Title: Cerebellar Stroke and Mood Disorders
Acronym: CERMOOD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CHUBX 2015/36
Record Dates: First submitted 2018-04-05; First posted 2018-05-03 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Stroke
Keywords: Stroke; Cerebellum; Depression; Anxiety; Mood; Magnetic resonance imaging (MRI)
MeSH Terms: conditions — Stroke; Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Post-stroke mood disorders evaluation (Experimental): Each patient will be assessed by a clinical evaluation, will have a standardized psychological evaluation, will perform a brain MRI and will be given a smartphone and an actimeter for a one-week period for the purpose of ecological evaluations.
  Interventions: Other: Post stroke mood disorders evaluation

INTERVENTIONS:
Other: Post stroke mood disorders evaluation — Each patient will be assessed by a clinical evaluation, will have a standardized psychological evaluation, will perform a brain MRI and will be given a smartphone and an actimeter for a one-week period for the purpose of ecological evaluations

SUMMARY:
Post-stroke mood disorders (PSMD), including depression, anxiety and apathy, are observed in about 30 % of stroke patients at follow-up 3 or 4 months after stroke occurrence. They impair the functional outcome of the patients and their quality of life. Among the different brain structures involved in PSMD the role of the cerebellum has been under-evaluated while it is now well-known to be involved in mood regulation. The aim of this study will be to describe the characteristics of early and late mood disorders following a first acute ischemic cerebellar stroke using face to face interviews and mobile technologies and investigate their pathophysiological mechanisms through advanced brain Magnetic resonance imaging (MRI) evaluation of cortico-cerebello-cortical morphological and functional connectivity.

DETAILED DESCRIPTION:
Stroke is the leading cause of acquired disability in adults. Beyond these physical consequences, stroke is a major cause of mood disorders (depression, anxiety, apathy), affecting more than 30% of patients at 3 months after the initial accident. These mood disorders impair patient's quality of life and their post-stroke functional recovery. Their detection is usually based on an interview conducted during a follow-up visit and intensity is measured through dedicated scales. However the sensitivity of these assessments could be improved by multiple daily ecological assessments carried out in the patient environment through mobile technologies such as smartphones (Experience Sampling Method) and actimeters. Moreover, a better understanding of the pathophysiological mechanisms underlying the presence of post-stroke mood disorders could improve their management. Clinical factors such as the severity of the disability or the female gender are associated with the occurrence of mood disorders but the independent role of the anatomical location of brain injury remains uncertain. During the last decade many studies have suggested the role of the cerebellum in the regulation of cognition and, to a lesser extent, mood. An anatomical or functional impairment of the cortico-cerebellar-cortical loops might contribute to the occurrence of the mood disorders observed in some patients with cerebellar lesion.

The aim of this project is to explore in the context of a cerebellar infarct the transverse association between the presence of post-stroke mood disorders, detected both by standard evaluations and assessments conducted in the ecological environment, and the functional and structural alteration of cortico-cerebellar-cortical loops evaluated by MRI.

ELIGIBILITY:
Inclusion Criteria :

* Patients with a first ischemic stroke affecting the cerebellum and returning to a post-visit AVS at 4 ± 1 month
* Age > 18 ans
* Modified Rankin Scale pre-stroke ≤ 1

Exclusion Criteria :

* History of central neurological disorder
* Pre-stroke cognitive impairment (IQ-code> 3.3) or post-stroke cognitive disorder defined by a MoCA < 24
* History of mood disorders history in the 6 months prior stroke (clinical screening)
* Moderate to severe leukoencephalopathy (Fazekas score ≥ 2 )
* Unable to use a smartphone (aphasia, visual disorder…)
* Participation in a pharmacological protocol involving psychotropic drugs (anxiolytics, antidepressants, antipsychotics) or a non-pharmacological protocol involving psychotherapeutic management
* Pregnancy
* MRI contra-indication(pacemaker, claustrophobia ...)
* Non affiliated to the French social insurance

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-01-16 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Center of Epidemiological Studies-Depression scale (CES-D) | Day 0
  Evaluation of depressive syndrome defined by a score> 17 for men and> 23 for women according to the CES-D
Beck Anxiety Inventory (BAI) | Day 0
  Evaluation of anxiety disorder defined by a score> 22 on the BAI scale
Apathy Inventory (AI) | Day 0
  Apathetic syndrome defined by a score > 2 on AI.

SECONDARY OUTCOMES:
Experience Sampling Method (ESM) evaluations | During 7 days
  Evaluation of daily-life mood disorders using one-week Experience Sampling Method (ESM) evaluations (smartphone)
Actimetry | During 7 days
  Circadian rhythms : sleep fragmentation and relative amplitude of circadian rhythms measured using one-week actimetry.
Trait-Meta-Mood-Scale (TMMS) | Day 0
  Evaluation of emotional dysregulation
Trait-Meta-Mood-Scale (TMMS) | 24 to 48 months
  Evaluation of emotional dysregulation
Interpersonal Reactivity Index (IRI) | Day 0
  Evaluation of emotional dysregulation
Interpersonal Reactivity Index (IRI) | 24 to 48 months
  Evaluation of emotional dysregulation
Facial emotion recognition tests | Day 0
  Evaluation of emotional dysregulation
Facial emotion recognition tests | 24 to 48 months
  Evaluation of emotional dysregulation
Brain Magnetic Resonance Imaging | Day 0
  Indexes of the structural and functional integrity of emotional regulation networks
Center of Epidemiological Studies-Depression scale (CES-D) | 24 to 48 months
  Evaluation of depressive syndrome defined by a score> 17 for men and> 23 for women according to the CES-D
Beck Anxiety Inventory (BAI) | 24 to 48 months
  Evaluation of anxiety disorder defined by a score> 22 on the BAI scale
Apathy Inventory (AI) | 24 to 48 months
  Apathetic syndrome defined by a score > 2 on AI.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Bordeaux, Bordeaux, France